CLINICAL TRIAL: NCT03399240
Title: Clinical Evaluation of the Accuracy of Vitastiq Device for Tracking Vitamin and Mineral Trend in Human Body
Acronym: VITASTIQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitastiq d.o.o. (Industry)
Collaborators: MEDEDUS, Ljubljana, Slovenia (Unknown); Adria Lab, Ljubljana, Slovenia (Unknown); Vizera d.o.o. (Industry); Faculty of Pharmacy, Ljubljana, Slovenia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Vita-01
Record Dates: First submitted 2018-01-05; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: No Conditions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitastiq device (Experimental): Vitastiq device is used for about 2 months to perform Vitastiq readings every day, preferably in the morning.
  Interventions: Device: Vitasitiq device

INTERVENTIONS:
Device: Vitasitiq device — Participant uses Vitastiq device for about 2 months to perform Vitastiq readings every day, preferably in the morning. On day 1, 29 and 57 participants' blood sampling is collected and analysed, and measurements using Vitastiq device are performed.

SUMMARY:
This is a single site evaluation study of Vitastiq device accuracy in healthy men and women in ratio 1:1 (approximately) aged between 18 and 64 years. A total of 45 Vitastiq personal devices will be used by volunteers for two months. The Vitastiq device will be evaluated during three site visits: on day 1, 29 ± 4 days and 57 ± 4 days. During site visit days, blood sampling will be collected and analysed and readings using Vitastiq device will be performed. Data will be analysed retrospectively to evaluate Vitastiq performance compared to blood tests results.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form (ICF) is signed by a volunteer
* Age between 18 and 64 years at the time of the signature of ICF
* A body mass index (BMI) between 18 and 28 kg/m2
* Healthy, meaning absence of any chronic or acute medical therapy for a month prior to the inclusion to the study
* Willing to follow all study procedures, including attending all site visits, and keeping a food diary and diary of activities on a weekly basis

Exclusion Criteria:

* Intake of any drugs to treat chronic disease within 1 month before the beginning and during the study
* Intake of any drugs to treat serious acute disease within 1 month before the beginning of the study and within 5 days of each visit
* Any clinically significant medical history of serious digestive tract, liver, kidney, skin or haematological disease or hormone imbalance
* Pregnant and breastfeeding women
* Women who planning pregnancy during the study
* Inadequate veins (in the opinion of the investigator)
* Known drug or alcohol abuse
* Using any form of nicotine or tobacco
* Mental incapacity that precludes adequate understanding or cooperation
* Participation in another investigational study or blood donation within 3 months prior to or during this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Vitastiq device accuracy and performance | 30 minutes
  Vitastiq accuracy performance is at least 70% meaning that at least 70% of Vitastiq readings for each mineral and vitamin fall within the range of matching blood test results.

SECONDARY OUTCOMES:
Vitastiq readings method is repeatable | 30 minutes
  Vitastiq readings method is at least 80% repeatable. It means that at least 80% of Vitastiq readings for each mineral and vitamin performed by investigators and participant in the time frame of 30 minutes are comparable.

CONTACTS AND LOCATIONS:
Locations (1):
- Adria Lab d.o.o., Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03399240/Prot_SAP_000.pdf